CLINICAL TRIAL: NCT05966662
Title: Prospective, Multicenter, Single-Arm IDE Study of the Shockwave Coronary Intravascular Lithotripsy (IVL) System With the Shockwave C2+ 2Hz Coronary IVL Catheter in Calcified Coronary Arteries (Disrupt CAD Duo Study)
Brief Title: Shockwave C2+ 2Hz Coronary IVL Catheter in Calcified Coronary Arteries (Disrupt CAD DUO)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 68277
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Intravasular Lithotripsy; PCI
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Shockwave C2+ 2Hz Coronary IVL Catheter with Shockwave Intravascular Lithotripsy (IVL) System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single-Arm (Experimental): Subjects with de novo, calcified coronary artery lesions presenting with stable, unstable, or silent ischemia that are suitable for percutaneous coronary intervention (PCI).
  Interventions: Device: IVL with Shockwave C2+ 2Hz Coronary IVL Catheter

INTERVENTIONS:
Device: IVL with Shockwave C2+ 2Hz Coronary IVL Catheter — Lithotripsy-enabled, low-pressure balloon dilatation of severely calcified, stenotic de novo coronary arteries prior to stenting.

SUMMARY:
This investigational device exemption (IDE) study is to assess the safety and effectiveness of the Shockwave Coronary Intravascular Lithotripsy (IVL) System with the Shockwave C2+ 2Hz Coronary IVL Catheter to treat de novo, calcified, stenotic, coronary lesions prior to stenting.

DETAILED DESCRIPTION:
The Shockwave Coronary Intravascular Lithotripsy (IVL) System with the Shockwave C2+ 2Hz Coronary IVL Catheter is indicated for lithotripsy-enabled, low-pressure balloon dilatation of severely calcified, stenotic de novo coronary arteries prior to stenting.

Up to 145 subjects (138 evaluable) subjects with de novo, calcified coronary artery lesions presenting with stable, unstable, or silent ischemia that are suitable for percutaneous coronary intervention (PCI) will be enrolled at up to 20 US sites.

Enrollment duration will be approximately 10-12 months and study duration will be approximately 2 years.

Each subject will be followed through discharge, 30 days, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:Subjects are required to meet all of the following inclusion criteria in order to be enrolled in the clinical study.

General Inclusion Criteria

1. Subject is ≥18 years of age
2. Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for PCI
3. For subjects with unstable ischemic heart disease, biomarkers (CK-MB and troponin) must be less than or equal to the upper limit of the laboratory normal within 12 hours prior to the procedure (note: both must be normal)
4. For subjects with stable ischemic heart disease, biomarkers may be drawn prior to the procedure or at the time of the procedure from the side port of the sheath

   1. If drawn prior to the procedure, biomarkers (CK-MB and troponin) must be less than or equal to the upper limit of the laboratory normal within 12 hours of the procedure (note: both must be normal)
   2. If drawn at the time of the procedure from the side port of the sheath prior to any intervention, biomarker results do not need to be analyzed prior to enrollment
5. Left ventricular ejection fraction >25% within 6 months (note: in the case of multiple assessments of LVEF, the measurement closest to enrollment will be used for this criterion; may be assessed at time of index procedure)
6. Subject or legally authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures
7. Non-target lesions requiring PCI may be treated either

   1. >30 days prior to the study procedure if the procedure was unsuccessful or complicated; or
   2. >24 hours prior to the study procedure if the procedure was successful and uncomplicated (defined as a final lesion angiographic diameter stenosis <30% and TIMI 3 flow (visually assessed) for all non-target lesions and vessels without perforation, cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation, and with no post-procedure biomarker elevation >normal; or
   3. >30 days after the study procedure

   Angiographic Inclusion Criteria
8. The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure
9. Single de novo target lesion stenosis of protected LMCA, or LAD, RCA or LCX (or of their branches) with

   1. Stenosis of ≥70% and <100%, or
   2. Stenosis ≥50% and <70% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve value ≤0.80, or iFR <0.90 or IVUS or OCT minimum lumen area ≤4.0 mm2
10. The target vessel reference diameter must be ≥2.5 mm and ≤4.0 mm
11. The lesion length must not exceed 40 mm
12. The target vessel must have TIMI flow 3 at baseline (visually assessed; may be assessed after pre- dilatation)
13. Evidence of calcification at the lesion site by, a) angiography, with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion, OR by b) IVUS or OCT, with presence of ≥270 degrees of calcium on at least 1 cross section
14. Ability to pass a 0.014" guide wire across the lesion

Exclusion Criteria: Subjects who meet any of the following exclusion criteria may not be enrolled in the study:

General Exclusion Criteria

1. Any comorbidity or condition which may reduce compliance with this protocol, including follow-up visits
2. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint
3. Subject is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrollment)
4. Unable to tolerate antiplatelet/anticoagulation therapy per society guidelines
5. Subject has an allergy to imaging contrast media which cannot be adequately pre-medicated
6. Subject experienced an acute MI (STEMI or non-STEMI) within 30 days prior to index procedure, defined as a clinical syndrome consistent with an acute coronary syndrome with troponin greater than 1 times the local laboratory's upper limit of normal
7. New York Heart Association (NYHA) class III or IV heart failure
8. Subject has acute or chronic renal disease with eGFR <30 ml/min/1.73m2 (using CKD-EPI formula)
9. History of a stroke or transient ischemic attack (TIA) within 60 days, or any prior intracranial hemorrhage or permanent neurologic deficit
10. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 3 months
11. Untreated pre-procedural hemoglobin <10 g/dL or intention to refuse blood transfusions if one should become necessary
12. Coagulopathy, including but not limited to platelet count <100,000 or International Normalized ratio (INR) > 1.7 (INR is only required in subjects who have taken warfarin within 2 weeks of enrollment)
13. Subject has a hypercoagulable disorder such as polycythemia vera, platelet count >750,000 or other related blood disorders
14. Subject has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics
15. Subjects with clinical evidence of cardiogenic shock
16. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
17. Subjects with a life expectancy of less than 1 year
18. Non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days prior to the index procedure
19. Planned non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days after the index procedure
20. Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
21. Planned use of atherectomy, scoring or cutting balloon, or any investigational device other than lithotripsy

    Angiographic Exclusion Criteria
22. Unprotected left main diameter stenosis >30%
23. Definite or possible thrombus (by angiography or intravascular imaging) in the target vessel
24. Evidence of aneurysm in target vessel within 10 mm of the target lesion
25. Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft
26. Previous stent within 5 mm of the target lesion regardless of the timing of its implantation
27. Angiographic evidence of a dissection or perforation in the target vessel at baseline or after guidewire passage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Heart Center Research, Huntsville, Alabama
  - Scripps Clinic, La Jolla, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Health, Hollywood, Florida
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Loyola University, Chicago, Illinois
  - Norton Heart and Vascular Institute, Louisville, Kentucky
  - Essentia Health St. Mary's Heart & Vascular Center, Duluth, Minnesota
  - Washington University, St Louis, Missouri
  - Northwell Health/Lenox Hill, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - The Christ Hospital, Cincinnati, Ohio
  - UPMC Pinnacle Health, Harrisburg, Pennsylvania
  - WellSpan Health - York, York, Pennsylvania
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Methodist Hospital, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent to Treat: Data analyzed from all enrolled participants through 30 days.
Period: Overall Study
Arm/Group | Intent to Treat
Started | 145
Completed | 145
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single-Arm
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean | 70.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 134
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Black or African American | 9
  Native Hawaiian or Other Pacific Islander | 0
  White | 120
  Unknown/ Not specified | 1
  Other | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (6.4)
BMI Categories 1 [Count of Participants; unit: Participants] — NIH BMI categories: underweight=BMI below 18.5; healthy weight=BMI of 18.5 to 24.9; overweight=BMI of 25 to 29.9; obesity=BMI of 30 or above
  Participants
    Underweight | 1
    Healthy weight | 33
    Overweight | 55
    Obesity | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Freedom From Major Adverse Cardiac Events (MACE) Within 30 Days Post-procedure
Description: Freedom from MACE within 30 days of the index procedure. MACE is defined as a composite occurrence of: cardiac death, myocardial infarction (MI), target vessel revascularization (TVR) after the completion of the index procedure.
Time Frame: within 30 days of index procedure
Population: One (1) subject experienced device delivery failure and was not included in the analysis.
Measure: Number; unit: Percentage of participants
Groups:
- Intent to Treat: Data on enrolled participants was collected through 30-days for primary endpoints.
Arm/Group | Intent to Treat
Number analyzed (Participants) | 144
Percentage of participants | 98.6

2. Primary Outcome: Percentage of Participants With Procedural Success (Residual Stenosis ≤30%)
Description: Procedural Success post stent delivery with a residual stenosis ≤30% (core laboratory assessed) and without in-hospital MACE.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 6 hours post procedure
Population: One (1) participant was not treated with the C2+ 2Hz catheter. Of those treated, one did not receive a stent during the index procedure and was not included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 143
Percentage of participants | 97.9

3. Secondary Outcome: Number of Participants With Device Crossing Success
Description: Device Crossing Success is defined as the ability to deliver the IVL catheter across the target lesion, and delivery of lithotripsy without serious angiographic complications immediately after IVL.
Time Frame: at the end of procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intent to Treat: Data on enrolled participants was collected through 30-days for secondary endpoints.
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Participants | 143

4. Secondary Outcome: Number of Participants With Angiographic Success (Residual Stenosis <50%)
Description: Angiographic Success defined as stent delivery with <50% residual stenosis and without serious angiographic complications.
Time Frame: at the end of procedure
Population: One (1) participant was not included as they were missing final angiographic images for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 144
Participants | 140

5. Secondary Outcome: Number of Participants With Procedural Success (Residual Stenosis <50% and Without In-hospital MACE)
Description: Procedural Success defined as stent delivery with a residual stenosis <50% (core laboratory assessed) and without in-hospital MACE.
Time Frame: at the end of the procedure
Population: One (1) subject did not receive a stent during the index procedure and was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 144
Participants | 141

6. Secondary Outcome: Number of Participants With Angiographic Success (Residual Stenosis ≤30%)
Description: Angiographic Success defined as stent delivery with ≤30% residual stenosis and without serious angiographic complications.
Time Frame: at end of procedure
Population: One (1) participant was not included in the analysis as they were missing final angiographic images for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 144
Participants | 140

7. Secondary Outcome: Number of Participants With Serious Angiographic Complications
Description: Serious angiographic complications defined as severe dissection (Type D to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow.
Time Frame: at end of procedure
Population: One (1) subject was not included as they were missing final angiographic images for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 144
Participants | 0

8. Secondary Outcome: Target Lesion Failure Rate at 30 Days
Description: Target lesion failure (TLF)is defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or ischemia-driven target lesion revascularization (ID-TLR) by percutaneous or surgical methods. 30 day rates are presented as proportions.
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of participants | 0.7

9. Secondary Outcome: All-Cause Death Rate at 30 Days
Description: Percentage of participants who experienced death (all-cause) through 30 days post index procedure.
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of participants
Groups:
- Intent to Treat: Data on enrolled participants was collected through 30 days for secondary endpoints.
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of participants | 0

10. Secondary Outcome: Cardiac Death Rate at 30 Days
Description: Percentage of participants who experienced cardiac death through 30 days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of participants | 0

11. Secondary Outcome: MI Rate at 30 Days
Description: Percentage of participants who experienced myocardial infarction through 30 days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of participants | 0.7

12. Secondary Outcome: Target Vessel-MI (TV-MI) Rate at 30 Days
Description: Percentage of participants who experienced MI attributable to the target vessel through 30 days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of participants | 0.7

13. Secondary Outcome: Procedural MI Rate at 30 Days
Description: Percentage of participants who experienced procedural myocardial infarction through 30 days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 0.7

14. Secondary Outcome: Non-Procedural MI Rate at 30 Days
Description: Percentage of participants who experienced Non-Procedural MI defined as spontaneous MI beyond discharge (4th Universal Definition) through 30 days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of participants | 0

15. Secondary Outcome: Ischemia Driven-Target Vessel Revascularization (ID-TVR) Rate at 30 Days
Description: Percentage of participants who experienced a Ischemia-Driven Target Vessel Revascularization through 30-days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 0

16. Secondary Outcome: Ischemia-Driven Target Lesion Revascularization (ID-TLR) Rate at 30 Days
Description: Percentage of participants who experienced a Ischemia-Driven Target Lesion Revascularization through 30-days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 0

17. Secondary Outcome: Non-Ischemia-Driven Target Vessel Revascularization (Non-ID-TVR) Rate at 30 Days
Description: Percentage of participants who experienced a Non-Ischemia-Driven Target Vessel Revascularization through 30-days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 0

18. Secondary Outcome: Non-ID-TLR Rate at 30 Days
Description: Percentage of participants who experienced a Non-Ischemia-Driven Target Lesion Revascularization through 30-days post index procedure
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 0.7

19. Secondary Outcome: Any Revascularizations Rate at 30 Days
Description: Percentage of participants who experienced any revascularizations (ID and non-ID) through 30 days post index procedure.
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 4.1

20. Secondary Outcome: Stent Thrombosis Rate at 30 Days
Description: Percentage of participants who experienced any stent thrombosis (definite, probable, definite or probable) through 30 days post index procedure.
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 0

21. Secondary Outcome: Rate of MI Using the 4th Universal Definition at 30 Days
Description: Percentage of participants who experienced MI using the 4th Universal Definition through 30 days post index procedure.
Time Frame: within 30 days of index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 145
Percentage of Participants | 7.6

ADVERSE EVENTS:
Time Frame: 30 days
Description: All Adverse events were summarized overall for the Intent to Treat population through 30-days of index procedure.
Groups:
- Intent to Treat (ITT): Adverse Events through 30 Days including all cause mortality, serious adverse events and non-serious adverse events that exceeded a 2.5% threshold.
Arm/Group | Intent to Treat (ITT)
All-Cause Mortality (participants affected / at risk) | 0/145
Serious Adverse Events (participants affected / at risk) | 13/145
Other Adverse Events (participants affected / at risk) | 9/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent to Treat (ITT) (N=145)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) — Non-cardiac chest pain
Plaque shift (Injury, poisoning and procedural complications) | 2 (2)
Influenza virus test positive (Investigations) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent to Treat (ITT) (N=145)
Coronary artery dissection (Cardiac disorders) | 4 (4)
Plaque shift (Injury, poisoning and procedural complications) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is more than 45 days but less than or equal to 90 days from the date that the communication is submitted to the sponsor for review. The sponsor cannot unilaterally extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT05966662/Prot_SAP_000.pdf